CLINICAL TRIAL: NCT00215618
Title: Clinical Evaluation of Uterine Balloon Therapy System for Menorrhagia
Brief Title: Uterine Balloon Treatment for Heavy Period Bleeding.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: David Robinson MD, Ethicon Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-010
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Uterine Balloon Therapy with post procedure curettage
  Interventions: Device: Uterine Balloon Therapy
- 2 (Experimental): Uterine Balloon Therapy without post-procedure curettage
  Interventions: Device: Uterine Balloon Therapy

INTERVENTIONS:
Device: Uterine Balloon Therapy — UBT with post procedure curettage
  Other Names: with post procedure curettage
  Arms: 1
Device: Uterine Balloon Therapy — UBT without post procedure curettage
  Other Names: without post procedure curettage
  Arms: 2

SUMMARY:
The purpose of this research is to determine the proportion of women who achieve permanent cessation of bleeding after Uterine Balloon Therapy (UBT) for the treatment of heavy uterine bleeding.

DETAILED DESCRIPTION:
This study was also designed to determine the effect of a post procedure curettage on bleeding patterns and post-operative discharge and pain.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 30 years of age who is premenopausal and for whom childbearing is complete.
* Excessive menstrual bleeding documented by a diary score of at least 150.
* Have documented 3 months failed medical therapy or either a) contraindicated for or b) refused medical therapy.
* Have an anatomically normal uterine cavity sounding at least 4cm, but not greater than 12cm.
* Have a normal pap smear and no unexplained abnormal pap smears within 1 year of the procedure.
* Agree not to switch from hormonal to non-hormonal contraception or vice versa during or just prior to the study.
* Agree to use reliable contraception throughout the study.
* Freely agree to participate in the study, including all study related procedures and evaluations, and document this agreement by signing informed consent documentation.

Exclusion Criteria:

* Active pelvic inflammatory disease (PID) or recurrent chronic PID.
* Active genital or urinary tract infection at the time of the procedure.
* History of malignancy of the reproductive system within 5 years of the procedure or have ever had malignancy of the endometrium.
* Endometrial neoplasia, determined by endometrial biopsy taken within 6 months of procedure.
* Cavity distorting submucous myoma(s) determined by preoperative hysterogram, hysteroscopy, or transvaginal sonography within 6 months of the procedure.
* Previous endometrial ablation procedure.
* Previous uterine surgeries (such as full thickness myomectomy, subserosal myomectomy, uterine reconstruction, or any surgery in which thinning of the uterine musculature could occur) except for low transverse caesarean section.
* Pregnant or desirous of future pregnancy.
* Taken endometrial suppression medication, except for oral contraceptives, within 3 months of the procedure.
* Concurrent open or laparoscopic surgery.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-03; Primary Completion 2006-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Incidence of post-procedure amenorrhea in women treated with uterine balloon therapy. | 6 and 12 mo

SECONDARY OUTCOMES:
Post-procedure bleeding levels | 2 and 3 yrs
Effect of post-procedure curettage on bleeding patterns, post-operative discharge and post-operative pain. | 2 and 3 yrs
System utility as indicated by equipment events that require intervention. | perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Cash, MD, Principal Investigator — Oakwood Hospital and Medical Center

REFERENCES:
- [Derived] Cash C Jr, Garza-Leal J, Donovan A, Guidry C, Romanowski C, Patel B. Clinical evaluation of long-term safety and effectiveness of a third-generation thermal uterine balloon therapy system for heavy menstrual bleeding. J Minim Invasive Gynecol. 2012 Jul-Aug;19(4):469-76. doi: 10.1016/j.jmig.2012.03.015. PMID 22748952